CLINICAL TRIAL: NCT01605162
Title: Phase 2 Study of the Poly(ADP-Ribose) Polymerase Inhibitor E7016 in Combination With Temozolomide in Subjects With Wild Type BRAF Stage IV or Unresectable Stage III Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7016-A001-201
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Wild Type BRAF Stage IV Melanoma; Unresectable Stage III Melanoma
MeSH Terms: interventions — 10-((4-hydroxypiperidin-1-yl)methyl)chromeno(4,3,2-de)phthalazin-3(2H)-one

ARMS (1):
- E7016 plus TMZ (Experimental)
  Interventions: Drug: TMZ; Drug: E7016

INTERVENTIONS:
Drug: TMZ — TMZ (at 150 mg/m2) will be administered orally according to the instructions on the product label, on Days 1 through 5 of the same 28-day cycle as E7016. TMZ capsules should be taken immediately after E7016. No food or drink intake, except water, will be allowed for 2 hours before or after administration.
Drug: E7016 — E7016 capsules will be administered in the morning after at least a 2-hour fast. Subjects will be instructed not to eat or drink anything except water in the 2 hours prior and 2 hours after drug administration. Subjects will record the time at which they ate.
  For the Single-Dose PK Period, 320 mg of E7016 will be administered once on Day -2. For the Multiple-Dose Treatment Cycle(s), 320 mg E7016 will be administered QD on Days 1 through 7 of each 28-day cycle.

SUMMARY:
This is a Phase 2, open-label, multicenter study to assess the PFS-6m of E7016 at the selected dose of 320-mg once daily (QD) in combination with 150-mg/m2 of Temozolomide (TMZ) in subjects with wt BRAF Stage IV or unresectable Stage III melanoma with disease progression. Eligible subjects must have measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be included in this study:

1. Males and females greater than or equal to 18 years of age
2. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol
3. Life expectancy greater than or equal to 3 months after starting E7016
4. Performance status of 0 - 2 on the Eastern Cooperative Oncology Group (ECOG) scale
5. Histopathologically confirmed diagnosis of melanoma with wt BRAF status (except melanoma of intraocular origin) with disease progression
6. American Joint Committee on Cancer (AJCC) Stage IV melanoma or unresectable Stage III melanoma
7. Measurable disease meeting the following criteria:

   * At least one lesion of greater than or equal to 1.0 cm in the longest diameter for a non-lymph node or greater than or equal to 1.5 cm in the short-axis diameter for a lymph node which is serially measurable according to RECIST 1.1 using computerized tomography/magnetic resonance imaging (CT/MRI). If there is only one target lesion and it is a non-lymph node, it should have a longest diameter of greater than or equal to 1.5 cm.
   * Lesions that have had external beam radiotherapy (EBRT) or loco-regional therapies such as radiofrequency (RF) ablation must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion.
8. Subjects with brain metastases will be eligible under the following conditions:

   * have undergone complete surgical excision and are more than 1 month post-surgery with no radiographic evidence of disease recurrence in the brain or
   * have undergone stereotactic radio surgery (gamma knife procedure or radiotherapy ) and are more than 1 month post procedure and with no radiographic evidence of disease progression in the brain and
   * are asymptomatic and
   * discontinued corticosteroid treatment and/or anticonvulsive therapy at least 1 week prior to Cycle 1, Day 1
9. Adequate renal function indicated by serum creatinine less than 1.5 mg/dL or calculated creatinine clearance greter than 50 mL/minute per Cockroft Gault formula
10. Adequate bone marrow reserve:

    * Absolute neutrophil count (ANC) greater than or equal to 1500/mm^3 (greater than or equal to 1.5 x 10^3/mL)
    * Platelets greater than or equal to 100,000/mm^3 (without transfusion)
    * Hemoglobin greater than or equal to 10 g/dL (less than 10.0 g/dL acceptable if corrected by growth factor or transfusion)
11. Adequate liver function:

    * Bilirubin less than or equal to 1.5 x the upper limit of normal (ULN) except for unconjugated hyperbilirubinemia of Gilbert's syndrome
    * Alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) less than or equal to 3 times ULN (less than or equal to 5 x ULN if subject has liver metastases)
12. Left ventricular ejection fraction (LVEF) greater than 50% on echocardiography or multiple-gated acquisition (MUGA) scanning
13. Females must not be lactating or pregnant at screening or baseline (as documented by a negative beta-human chorionic gonadotropin [B-hCG] test with a minimum sensitivity of 25 IU/L or equivalent units of B-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (i.e., bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing). Females of childbearing potential must not have had unprotected sexual intercourse within 30 days prior to study entry and must agree to use a highly effective method of contraception (e.g., total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. If currently abstinent, the subject must agree to use a double-barrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
14. Male subjects must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must meet the criteria above (i.e., not of childbearing potential or practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation).

Exclusion Criteria:

Subjects with any one of the following will be excluded from this study:

1. Subjects with melanoma of intraocular origin
2. Leptomeningeal metastasis or brain metastasis except as for inclusion criteria number 8
3. Subjects taking medications which are either strong CYP inhibitors or inducers
4. Subjects with active malignancies except for wt BRAF Stage IV and unresectable Stage III melanoma, basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, adequately treated Stage I or II cancer from which the subject is currently in complete remission, or any other cancer from which the subject has been disease-free for 5 years
5. Prior treatment with a PARP inhibitor
6. Prior treatment with dacarbazine (DTIC) or TMZ containing regimens
7. Subjects with known allergy, hypersensitivity, or other contraindication to E7016, TMZ, or DTIC or any of the other components of the formulations
8. Subjects with known human immunodeficiency virus infection (HIV), active hepatitis B or C
9. Subjects with active infections requiring specific anti-infective therapy
10. Subjects who have had a major surgical procedure (including tumor resection) within 4 weeks prior to initiating E7016 treatment
11. Subjects scheduled for surgery during the projected course of the study
12. Chemotherapy, radiation therapy, or immunotherapy within 4 weeks prior to initiating E7016 treatment (6 weeks for mitomycin C or nitrosoureas) or any investigational agent within 30 days prior to the first dose of study drug or who have not recovered (Grade 0 or 1) from any acute toxicity related to previous anticancer treatment
13. Prolongation of QT corrected, the QT interval corrected for heart rate (QTc) interval (greater than 480 ms)
14. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II ; unstable angina; uncontrolled hypertension despite optimal treatment, myocardial infarction or stroke within 6 months of the first dose of study drug; or cardiac arrhythmia requiring medical treatment
15. Subjects with malabsorption syndrome or any other condition that might affect bioavailability of study drug (E7016 or TMZ)
16. Other relevant disease or adverse clinical conditions such as:

    * History of significant neurological (no neuropathy greater than Grade 2) or psychiatric disorders
    * Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis)
    * Significant non-neoplastic renal disease
    * Uncontrolled endocrine disease (e.g., diabetes mellitis, hypothyroidism or hyperthyroidism, adrenal disorder) i.e., requiring relevant changes in medication within the last month or hospital admission within the last 3 months
17. Any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in this study
18. Female who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The Progression Free Survival-6m rate defined as the proportion of subjects that are alive and progression-free at 6-months from the date of first dosing based on RECIST 1.1. | 6 months
  The Progression Free Survival-6m rate defined as the proportion of subjects that are alive and progression-free at 6-months from the date of first dosing based on RECIST 1.1. PFS-6m rate will be estimated from Kaplan-Meier (K-M) product-limit estimate of PFS.

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Services, Study Director — Eisai Inc.
Locations (1):
- Pittsburgh, Pennsylvania, United States